CLINICAL TRIAL: NCT06227442
Title: Predictor of Renal Involvement in Rheumatoid Arthritis:Value of Renal Resistive Index
Brief Title: Renal Resistive Index as a Predictor of Renal Involvement in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Noman Mohamed AbdElaziz, master, Assiut University
Other Study IDs: PORIIRA
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: will include 48 RA patients without renal affection.
  Interventions: Diagnostic Test: KDIGO criteria of 2010
- Group B: will include 48 RA patients with renal affection.
  Interventions: Diagnostic Test: KDIGO criteria of 2010
- Group C: will include 48 healthy control.
  Interventions: Diagnostic Test: KDIGO criteria of 2010

INTERVENTIONS:
Diagnostic Test: KDIGO criteria of 2010 — They are guidelines for the diagnosis, evaluation, and management of chronic kidney disease (CKD). They cover the classification of CKD stages based on glomerular filtration rate and albuminuria, criteria for diagnosing acute kidney injury, and recommendations for managing CKD-related complications.

SUMMARY:
Evaluation of resistive index on the renal artery as early predictor factor of renal affection in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disorder characterized by synovial hyperplasia and inflammation, progressive joint destruction, and significant disability (1). It can occur at any age, but it predominantly affects women, with a peak onset between the ages of 40 and 60. RA etiology is not yet clear, Recent studies have shown that its mechanism is closely related to genetics, environment, and immune response. Genes such as MHC and HLA-DR4 are involved in the occurrence of RA. (2) Renal complications in RA can range from mild abnormalities in kidney function to more severe conditions, such as glomerulonephritis and renal amyloidosis. Understanding these renal complications is crucial for healthcare providers to ensure comprehensive care for RA patients. (3.4) Vasculitis is an uncommon complication of RA (in approximately 2 to 5% of patients), males with RA are more likely (2 to 4 times more likely) than females with RA to develop RV. Rheumatoid vasculitis most often occur in people with at least 10 years of severe disease. Fortunately, recent reports have noted declines in the prevalence of RV ( 5.6). So The renal arterial resistive index (RI)which is a sonographic index of intrarenal arteries defined as (peak systolic velocity - end-diastolic velocity) / peak systolic velocity. The normal range is 0.50-0.70. Elevated values are associated with poorer prognosis in various renal disorders .

ELIGIBILITY:
Inclusion Criteria:

* Patients of rheumatoid arthritis è renal affection
* Patients of rheumatoid arthritis without renal affection
* Patients of rheumatoid arthritis on drugs (NSAIDs, DMARDS, methotrexate..).

Exclusion Criteria:

* Diabetic and hypertensive patients, patients with hepatitis B, C viruses or liver cell failure, patients with acute kidney injury, patients with another autoimmune disease as (SLE, sjogren disease, multiple sclerosis, patients with malignancy, patients on another drugs otherwise rheumatoid arthritis drugs).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Base on determining the main outcome variable, the estimated minimum required sample size is 144 cases (48 case in each group)
  The sample size was calculated using G*power software 3.1.9.7 based on following assumptions:
  Mean serum creatinine level in RA patients without renal affection compared to mean serum creatinine level RA patients with renal affection and control group.
  The Effect size is estimated to be 0.3. Main statistical test is one way ANOVA ,Alpha=0.05, power=90
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating predictive value of renal resistive index in detection of rheumatoid arthritis. | baseline
  Assesses the predictive utility of renal resistive index in detecting rheumatoid arthritis. Delve into the exploration of whether renal resistive index serves as a reliable marker, offering valuable insights into the potential diagnostic relevance for rheumatoid arthritis.

SECONDARY OUTCOMES:
Identify the risk factor for renal complication in RA patients | baseline
  Explore the factors contributing to renal complications in rheumatoid arthritis (RA) patients with a focus on identifying key risk factors. Uncover insights that enhance our understanding of the complex relationship between RA and renal involvement, ultimately aiding in targeted prevention and management strategies.

REFERENCES:
- [Background] Li XF, Sun YY, Bao J, Chen X, Li YH, Yang Y, Zhang L, Huang C, Wu BM, Meng XM, Li J. Functional role of PPAR-gamma on the proliferation and migration of fibroblast-like synoviocytes in rheumatoid arthritis. Sci Rep. 2017 Oct 4;7(1):12671. doi: 10.1038/s41598-017-12570-6. PMID 28978936
- [Background] Jung JY, Kim YB, Kim JW, Suh CH, Kim HA. Biologic therapy for amyloid A amyloidosis secondary to rheumatoid arthritis treated with interleukin 6 therapy: Case report and review of literature. Medicine (Baltimore). 2021 Aug 13;100(32):e26843. doi: 10.1097/MD.0000000000026843. PMID 34397890
- [Background] Oweis AO, Alawneh KM, Alshelleh SA, Alnaimat F, Alawneh D, Zahran DJ. Renal dysfunction among rheumatoid arthritis patients: A retrospective cohort study. Ann Med Surg (Lond). 2020 Nov 4;60:280-284. doi: 10.1016/j.amsu.2020.11.011. eCollection 2020 Dec. PMID 33204418
- [Background] Alamanos Y, Voulgari PV, Drosos AA. Incidence and prevalence of rheumatoid arthritis, based on the 1987 American College of Rheumatology criteria: a systematic review. Semin Arthritis Rheum. 2006 Dec;36(3):182-8. doi: 10.1016/j.semarthrit.2006.08.006. Epub 2006 Oct 11. PMID 17045630
- [Background] Vollertsen RS, Conn DL. Vasculitis associated with rheumatoid arthritis. Rheum Dis Clin North Am. 1990 May;16(2):445-61. PMID 2189161